CLINICAL TRIAL: NCT03516006
Title: Intra-arterial Injection of Umbilical Cord Mesenchymal Stem Cells in Primary Sclerosing Cholangitis
Brief Title: Umbilical Cord Mesenchymal Stem Cells in Primary Sclerosing Cholangitis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: Principal Investigator, Dongliang Li, Professor, Fuzhou General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCMSC-PSC
Record Dates: First submitted 2017-09-20; First posted 2018-05-04 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-04

CONDITIONS: Primary Sclerosing Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UCMSC (Experimental): infusion of aUCMSC and Ursodeoxycholic acid therapy
  Interventions: Drug: UCMSC; Drug: UDCA
- UDCA (Active Comparator): Ursodeoxycholic acid therapy 15mg/kg/d
  Interventions: Drug: UDCA

INTERVENTIONS:
Drug: UCMSC — infusion of aUCMSC at day 0, 7, 14, and 21
  Arms: UCMSC
Drug: UDCA — oral administration of ursodeoxycholic acid (UDCA) 15mg/kg/d

SUMMARY:
Primary sclerosing cholangitis (PSC) is an idiopathic condition with intrahepatic cholangitis and fibrosis, leading to multifocal bile duct stricture. Its main clinical manifestations are chronic cholestatic lesions and is deemed as autoimmune liver disease. PSC are immune abnormalities that occurs in patients with genetic susceptibility. No other pathogenesis is revealed yet. Ursodeoxycholic acid is used as an empirical treatment, and there is no approved drug or a acceptable treatment regimen. The disease often progresses to liver decompensation and requires liver transplantation. In recent years, the clinical application of stem cell therapy has seen many important advances. Stem cells are characterized with properties of multiple differentiation, repair of damaged tissue and immuno-modulation. This study aims to employ UCMSCs to treat PSC patients and observe its efficacy and safety, and to explore the possible therapeutic mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* progressive PSC
* willing to give consent

Exclusion Criteria:

* decompensated liver cirrhosis
* total serum bilirubin >5ULN
* refractory ascites
* serum creatinine >1.5mg/dL
* Cirrhotic nodules with malignant tendencies
* primary biliary cholangitis
* IgG4-associated sclerosing cholangitis
* non-PSC induced bile duct stones
* biliary tract trauma
* recurrent suppurative cholangitis
* neoplastic disease
* pancreatic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
adverse effects regarding UCMSC infusion | 1 year

SECONDARY OUTCOMES:
Pathological score of liver inflammation | 1 year
Changes of biliary lesions in magnetic resonance image | 1 year
  softening in stiffness of bile duct
alanine aminotransferase | 1 year